CLINICAL TRIAL: NCT05500092
Title: An Open Label, Randomized Study of Neoadjuvant Nivolumab and Chemotherapy, With or Without Sub-ablative Stereotactic Body Radiation Therapy, for Resectable Stage IIA to IIIB Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Penn State University (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13627; CA209-6K6 (Other: Bristol Myers Squibb (BMS))
Record Dates: First submitted 2022-07-15; First posted 2022-08-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Resectable Stage IIA to IIIB Non-small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab; Carboplatin; Cisplatin; Pemetrexed; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab + Platinum Doublet Chemotherapy (Active Comparator): All participants will receive platinum-based doublet chemotherapy (PDC) along with nivolumab for 3 cycles every 3 weeks. Carboplatinum (AUC=5) can be used instead of Cisplatin (75 mg/m2) from cycle 2 for Cisplatin induced neuro/oto/nephrotoxicity as long as the subject remains eligible for doublet chemotherapy. Participants with nonsquamous tumors will receive pemetrexed (500 mg/m2). Participants with squamous tumors will receive either docetaxel (75 mg/m2 on day 1) or gemcitabine (1000 mg/m2 on days 1, 8). Cycles will be every 3 weeks and a maximum of a 2 week delay will be permitted for resolution of toxicities.
  Interventions: Drug: Nivolumab; Drug: Platinum Doublet
- Nivolumab + Platinum Doublet Chemotherapy + SBRT (8gy x 3) (Experimental): SBRT will be delivered near the conclusion of cycle 1 with platinum-based doublet chemotherapy (PDC) along with nivolumab for 3 cycles every 3 weeks. The intent is to deliver SBRT on three consecutive days when the concentration of radiosensitizing chemotherapy agents in the subject's system is at a minimum, to minimize toxicity risks. It is expected that some subjects may not receive SBRT on three consecutive days due to machine breakdown, inclement weather, or other logistic issues. Subjects must not receive SBRT within 72 hours after a cisplatin or carboplatin infusion
  Interventions: Drug: Nivolumab; Radiation: (8gy x 3); Drug: Platinum Doublet

INTERVENTIONS:
Drug: Nivolumab — Patients randomized to the Nivolumab + Platinum Doublet Chemotherapy only arm will receive three cycles of nivolumab at a dose of 360 mg every three weeks along with a platinum-based chemotherapy doublet (cisplatin or carboplatin plus pemetrexed for adenocarcinoma, cisplatin or carboplatin plus docetaxel, paclitaxel, or gemcitabine for squamous NSCLC) with sub-ablative stereotactic radiation therapy (8 Gy x 3) directed at the primary lung tumor
Radiation: (8gy x 3) — sub-ablative stereotactic radiation therapy (8 Gy x 3) directed at the primary lung tumor
  Arms: Nivolumab + Platinum Doublet Chemotherapy + SBRT (8gy x 3)
Drug: Platinum Doublet — Standard of care doublet platinum therapy
  Other Names: Carboplatinum; Cisplatin; Pemetrexed; Docetaxel; Gemcitabine

SUMMARY:
An open label, randomized study of neoadjuvant nivolumab and chemotherapy, with or without sub-ablative stereotactic body radiation therapy, for resectable stage IIA to IIIB non-small cell lung cancer

DETAILED DESCRIPTION:
Primary Objective

* To compare the complete pathological response rate after 3 cycles of neoadjuvant nivolumab and platinum-based doublet chemotherapy vs. the same regimen with the addition of sub-ablative stereotactic radiation therapy (8 Gy x 3) directed at the primary lung tumor.

Secondary Objectives

* To characterize the rate of Major Pathological Response (MPR), defined as ≤ 10% residual viable tumor cells at the time of surgical resection in the primary tumor and lymph nodes, as assessed by local pathology laboratory.
* To characterize rates of Event Free Survival (EFS), defined as survival without documented disease progression per RECIST v1.1 that precludes surgery for local or distant disease recurrence.

Exploratory Objectives

* To characterize the rate of pathological downstaging of biopsy confirmed positive lymph nodes not in the stereotactic body radiation therapy (SBRT) field.
* To characterize rates of Disease-Free Survival (DFS), defined as survival without local or distant recurrence or occurrence of new primary NSCLC.
* To characterize rates of Overall Survival (OS) after study enrollment.
* To characterize the incidence of adverse events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
* To describe surgical safety and the incidence and severity of surgery-related adverse events.
* To characterize rates of clearance of circulating tumor DNA (ctDNA) following neoadjuvant therapy and definitive surgical treatment
* To evaluate whole tumor RNA-sequencing (RNAseq) from pre- and post- treatment tissue samples to assess for predictors and signatures of pathologic response.
* To evaluate of gene expression in pre- and post-treatment blood samples to assess for predictors and signatures of complete pathologic response.
* To assess the expression characteristics of PD-L1, infiltrating immune cells and tumor mutational burden (TMB), and their association with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically proven clinical stages IIA (tumors > 4 cm), IIB, IIIA, and IIIB (T3 or T4, N2) NSCLC (AJCC version 8) and is considered eligible for surgical resection with curative intent. Patients with 2 primary non-small cell lung cancers are allowed.
2. Measurable disease, as defined by RECIST v1.1.
3. Parenchymal lung tumor deemed to be amenable to treatment with sub-ablative stereotactic body radiation therapy, as determined by a co-investigator from Radiation Oncology
4. Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) obtained from the subject prior to performing any protocol-related procedures.
5. Age > 18 years at time of study entry
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * Aspartate aminotransferase (SGOT)/Alanine Aminotransferase (SGPT), and alkaline phosphatase ≤ 2.5 x institutional upper limit of normal (ULN).
   * Serum creatinine clearance>50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (CL):

   Males:

   Creatinine CL (mL/min)

   = Weight (kg) x (140 - Age) . 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min)

   = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
8. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

   Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. No prior therapy for their lung cancer.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an investigational product during the last 3 weeks.
2. Active other primary malignancy excepting:

   * Malignancy treated with curative intent and with no known active disease and of low potential risk for recurrence.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ, in-situ urinary bladder cancer, treated localized prostate cancer and ductal carcinoma-in situ.
3. Current or prior use of immunosuppressive medication within 14 days before the first dose of nivolumab, with the exceptions of intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection), corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, and steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Patients with Grade ≥2 neuropathy.
5. Previous receipt of immunotherapy.
6. Active or prior documented autoimmune or inflammatory disorders that has required systemic treatment in the past year (including inflammatory bowel disease [e.g., colitis or Crohn's disease systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). No active diverticulitis within the previous 3 months. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
7. History of allogeneic organ transplant.
8. History of hypersensitivity to nivolumab or any excipient.
9. Uncontrolled intercurrent illness that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
10. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), active hepatitis B (known positive Hepatitis B virus surface antigen (HBsAg) result), active hepatitis C.
11. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of nivolumab monotherapy.
12. History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonitis (including drug induced), or evidence of active pneumonitis on screening chest CT scan.
13. Receipt of the last dose of therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, or other investigational agent) for an accepted other malignancy as defined in Section 3.3.2 within 30 days prior to the first dose of study drug for lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Complete Pathological Response Rate | After 3 cycles. Each cycle is defined as 3 weeks
  Complete pathological response (CPR) rate observed after neoadjuvant therapy and surgical resection. Complete pathological response will be defined as the absence of tumor cells in the resected specimen upon histopathological examination. CPR rate will be reported as a percentage along with a 95% Confidence Interval for each study arm.

SECONDARY OUTCOMES:
Major Pathological Response | After 3 cycles. Each cycle is defined as 3 weeks
  Major Pathological Response (MPR) rate will be assessed. MPR will be defined as ≤ 10% residual viable tumor cells, at the time of surgical resection, in the primary tumor and resected lymph nodes, as assessed by local pathology laboratory. MPR rate and corresponding 95% Clopper-Pearson confidence intervals will be calculated for each treatment arm.
Event Free Survival | From the time of enrollment up to approximately 5 years
  Event free survival (EFS) will be defined as survival without evidence of documented disease progression, per RECIST v1.1 criteria, that precludes surgery for local or distant disease recurrence. Results will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Brendon Stiles, MD, Principal Investigator — Montefiore Medical Center
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - Montefiore Medical Center-Albert Einstein College of Medicine, The Bronx, New York
  - White Plains Hospital (WPH), White Plains, New York
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No